CLINICAL TRIAL: NCT03241797
Title: Evaluation of EUS-guided FNA for Diagnosing Autoimmune Pancreatitis: a Prospective, Single-center Study
Brief Title: Evaluation of EUS-guided FNA for Diagnosing Autoimmune Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bin Cheng (Other)
Responsible Party: Sponsor-Investigator, Bin Cheng, professor, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AIP
Record Dates: First submitted 2017-07-29; First posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Autoimmune Pancreatitis
Keywords: AIP; EUS-FNA
MeSH Terms: conditions — Autoimmune Pancreatitis | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients who suggested having AIP (Experimental): Patients who suggested having AIP and underwent EUS-FNA biopsy by using a standard 22-gauge aspiration needle were enrolled between January 2013 and May 2017.
  Interventions: Procedure: EUS-FNA

INTERVENTIONS:
Procedure: EUS-FNA — Once the lesion was evaluated by EUS, the echoendoscopist would select the shortest pathway, while avoiding blood vessels, to reach the lesion. Under real-time visualization, slow-pull technique and suction technique were used to punctured each lesions. The specimens were expelled onto glass slides, and then prepared for histological and cytological examinations.

SUMMARY:
The aim is to evaluate EUS-FNA efficacy for AIP diagnosis using a 22-gauge (G) needle.

DETAILED DESCRIPTION:
Patients who suggested having Autoimmune pancreatitis (AIP) and underwent endoscopic ultrasound-guided fine needle aspiration (EUS-FNA） by using a standard 22-gauge aspiration needle were enrolled between January 2013 and May 2017. The enrollment criteria included age greater than 20 years at the time of enrollment; presence of imaging characteristics of AIP, as specified in the International Consensus Diagnostic Criteria（ICDC） (diffuse or segmental/focal enlargement with delayed enhancement and diffuse or segmental/focal or multiple irregular narrowing of the main pancreatic duct without marked upstream dilatation) was confirmed by computed tomography (CT), magnetic resonance imaging (MRI), or EUS. The exclusion criteria were steroid administration within 3 months before the initiation of treatment; refusal or inability to provide informed consent; episode of acute pancreatitis in previous 2 weeks; inability to safely perform EUS-FNA, such as cardiorespiratory dysfunction, mental diseases, coagulopathy and drug addiction.All procedures were performed under deep sedation by a single experienced endosonographer who had performed more than 500 cases. EUS-FNA was performed by using Olympus linear echoendoscopes , Diagnostic Ultrasound System and 22-G needle . Once the lesion was evaluated by EUS, the echoendoscopist would select the shortest pathway, while avoiding blood vessels, to reach the lesion. Under real-time visualization, slow-pull technique and suction technique were used to punctured each lesions. The specimens were expelled onto glass slides, and then prepared for histological and cytological examinations. Because neither pathologists nor cytologists were present on-site at our institution, the puncture was repeated until a whitish material could be observed macroscopically.Tissue samples were fixed in formalin and embedded in paraffin. A paraffin block was thin cut into serial sections and stained with hematoxylin-eosin(H&E). To detect infiltrated plasma cells, anti-IgG4 antibody would be done if necessary. The histologic analysis was made by an experienced pathologist who was blind to the kinds of studies referring to the histological criteria of the ICDC. The Lymphoplasmacytic sclerosing pancreatitis (LPSP ) findings are as follow: (1) Periductal lymphoplasmacytic infiltrate without granulocytic infiltration; (2) Obliterative phlebitis; (3)Storiform fibrosis; (4) Abundant (>10cells/HPF) immunoglobulin G4 (IgG 4)positive cells. The level-1 criteria of LPSP were positive for 3 or more of the 4 LPSP findings, and the level-2 criteria were positive for 2 of the 4 items. The idiopathic duct-centric chronic pancreatitis (IDCP) findings are as follow: (1) Granulocytic infiltration of duct wall (GEL) with or without granulocytic acinar inflammation; (2)Granulocytic and lymphoplasmacytic acinar infiltrate; (3)Absent or scant (0-10 cells/ High-power fields) IgG4-positive cells. The level-1 criteria of IDCP were positive for items (1) and (3), and the level-2 criteria were positive for items (2) and (3).Statistical analyses were performed with Statistical Analysis System (SAS) version 9.2. All tests were 2-tailed and a P value of less than 0.05 was considered to indicate a statistically significant difference. All category variables will be described in terms of the count and percentage using the χ 2 test, whereas the continuous variables will be described as mean ± standard deviation using τ tests or Wilcoxon rank-sum tests. Outpatients were observed for immediate complications in the recovery room for 2 hours and followed up on the day after the procedure to monitor for possible complications.

ELIGIBILITY:
Inclusion Criteria:

* age >20 years old, <85 years old ; probable AIP.

Exclusion Criteria:

* steroid administration within 3 months before the initiation of treatment; refusal or inability to provide informed consent; acute pancreatitis in previous 2 weeks; cardiorespiratory dysfunction; mental diseases; coagulopathy; drug addiction(asprin, clopidogrel).

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
evaluate the diagnostic yield of AIP patients by EUS-FNA . | 52 months
  The primary outcome measure is to evaluate the usefulness of EUS-FNA with 22-Gauge (G) needle in histological diagnosis of AIP patients.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Cheng, Doctor, Principal Investigator — Tongji Hospital; Yun Wang, Doctor, Study Chair — Tongji Hospital; Li Cao, Doctor, Study Director — Tongji Hospital
Locations (1):
- Tongji hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] SARLES H, SARLES JC, MURATORE R, GUIEN C. Chronic inflammatory sclerosis of the pancreas--an autonomous pancreatic disease? Am J Dig Dis. 1961 Jul;6:688-98. doi: 10.1007/BF02232341. No abstract available. PMID 13746542
- [Result] Hart PA, Kamisawa T, Brugge WR, Chung JB, Culver EL, Czako L, Frulloni L, Go VL, Gress TM, Kim MH, Kawa S, Lee KT, Lerch MM, Liao WC, Lohr M, Okazaki K, Ryu JK, Schleinitz N, Shimizu K, Shimosegawa T, Soetikno R, Webster G, Yadav D, Zen Y, Chari ST. Long-term outcomes of autoimmune pancreatitis: a multicentre, international analysis. Gut. 2013 Dec;62(12):1771-6. doi: 10.1136/gutjnl-2012-303617. Epub 2012 Dec 11. PMID 23232048
- [Result] Meng Q, Xin L, Liu W, Lin H, Tian B, Wang L, Li Z. Diagnosis and Treatment of Autoimmune Pancreatitis in China: A Systematic Review. PLoS One. 2015 Jun 25;10(6):e0130466. doi: 10.1371/journal.pone.0130466. eCollection 2015. PMID 26110658
- [Result] Hoki N, Mizuno N, Sawaki A, Tajika M, Takayama R, Shimizu Y, Bhatia V, Yamao K. Diagnosis of autoimmune pancreatitis using endoscopic ultrasonography. J Gastroenterol. 2009;44(2):154-9. doi: 10.1007/s00535-008-2294-2. Epub 2009 Feb 13. PMID 19214678
- [Result] Pearson RK, Longnecker DS, Chari ST, Smyrk TC, Okazaki K, Frulloni L, Cavallini G. Controversies in clinical pancreatology: autoimmune pancreatitis: does it exist? Pancreas. 2003 Jul;27(1):1-13. doi: 10.1097/00006676-200307000-00001. No abstract available. PMID 12826899
- [Result] Kim KP, Kim MH, Kim JC, Lee SS, Seo DW, Lee SK. Diagnostic criteria for autoimmune chronic pancreatitis revisited. World J Gastroenterol. 2006 Apr 28;12(16):2487-96. doi: 10.3748/wjg.v12.i16.2487. PMID 16688792
- [Result] Kim MH, Kwon S. Diagnostic criteria for autoimmune chronic pancreatitis. J Gastroenterol. 2007 May;42 Suppl 18:42-9. doi: 10.1007/s00535-007-2050-z. PMID 17520223
- [Result] Levy MJ, Reddy RP, Wiersema MJ, Smyrk TC, Clain JE, Harewood GC, Pearson RK, Rajan E, Topazian MD, Yusuf TE, Chari ST, Petersen BT. EUS-guided trucut biopsy in establishing autoimmune pancreatitis as the cause of obstructive jaundice. Gastrointest Endosc. 2005 Mar;61(3):467-72. doi: 10.1016/s0016-5107(04)02802-0. PMID 15758927
- [Result] Ishikawa T, Itoh A, Kawashima H, Ohno E, Matsubara H, Itoh Y, Nakamura Y, Nakamura M, Miyahara R, Hayashi K, Ishigami M, Katano Y, Ohmiya N, Goto H, Hirooka Y. Usefulness of EUS combined with contrast-enhancement in the differential diagnosis of malignant versus benign and preoperative localization of pancreatic endocrine tumors. Gastrointest Endosc. 2010 May;71(6):951-9. doi: 10.1016/j.gie.2009.12.023. PMID 20438884
- [Result] Iwashita T, Yasuda I, Doi S, Ando N, Nakashima M, Adachi S, Hirose Y, Mukai T, Iwata K, Tomita E, Itoi T, Moriwaki H. Use of samples from endoscopic ultrasound-guided 19-gauge fine-needle aspiration in diagnosis of autoimmune pancreatitis. Clin Gastroenterol Hepatol. 2012 Mar;10(3):316-22. doi: 10.1016/j.cgh.2011.09.032. Epub 2011 Oct 20. PMID 22019795
- [Result] Kanno A, Masamune A, Fujishima F, Iwashita T, Kodama Y, Katanuma A, Ohara H, Kitano M, Inoue H, Itoi T, Mizuno N, Miyakawa H, Mikata R, Irisawa A, Sato S, Notohara K, Shimosegawa T. Diagnosis of autoimmune pancreatitis by EUS-guided FNA using a 22-gauge needle: a prospective multicenter study. Gastrointest Endosc. 2016 Nov;84(5):797-804.e1. doi: 10.1016/j.gie.2016.03.1511. Epub 2016 Apr 9. PMID 27068878
- [Result] Kanno A, Ishida K, Hamada S, Fujishima F, Unno J, Kume K, Kikuta K, Hirota M, Masamune A, Satoh K, Notohara K, Shimosegawa T. Diagnosis of autoimmune pancreatitis by EUS-FNA by using a 22-gauge needle based on the International Consensus Diagnostic Criteria. Gastrointest Endosc. 2012 Sep;76(3):594-602. doi: 10.1016/j.gie.2012.05.014. PMID 22898417
- [Result] Yasuda I, Tsurumi H, Omar S, Iwashita T, Kojima Y, Yamada T, Sawada M, Takami T, Moriwaki H, Soehendra N. Endoscopic ultrasound-guided fine-needle aspiration biopsy for lymphadenopathy of unknown origin. Endoscopy. 2006 Sep;38(9):919-24. doi: 10.1055/s-2006-944665. PMID 16981110
- [Result] Iwashita T, Yasuda I, Tsurumi H, Goto N, Nakashima M, Doi S, Hirose Y, Takami T, Moriwaki H. Endoscopic ultrasound-guided fine needle aspiration biopsy for splenic tumor: a case series. Endoscopy. 2009 Feb;41(2):179-82. doi: 10.1055/s-0028-1119474. Epub 2009 Feb 12. PMID 19214901
- [Result] Mizuno N, Bhatia V, Hosoda W, Sawaki A, Hoki N, Hara K, Takagi T, Ko SB, Yatabe Y, Goto H, Yamao K. Histological diagnosis of autoimmune pancreatitis using EUS-guided trucut biopsy: a comparison study with EUS-FNA. J Gastroenterol. 2009;44(7):742-50. doi: 10.1007/s00535-009-0062-6. Epub 2009 May 12. PMID 19434362
- [Result] Na HK, Lee JH, Park YS, Ahn JY, Choi KS, Kim DH, Choi KD, Song HJ, Lee GH, Jung HY, Kim JH. Yields and Utility of Endoscopic Ultrasonography-Guided 19-Gauge Trucut Biopsy versus 22-Gauge Fine Needle Aspiration for Diagnosing Gastric Subepithelial Tumors. Clin Endosc. 2015 Mar;48(2):152-7. doi: 10.5946/ce.2015.48.2.152. Epub 2015 Mar 27. PMID 25844344
- [Result] Itoi T, Itokawa F, Kurihara T, Sofuni A, Tsuchiya T, Ishii K, Tsuji S, Ikeuchi N, Kawai T, Moriyasu F. Experimental endoscopy: objective evaluation of EUS needles. Gastrointest Endosc. 2009 Mar;69(3 Pt 1):509-16. doi: 10.1016/j.gie.2008.07.017. PMID 19231491
- [Result] Levy MJ, Wiersema MJ, Chari ST. Chronic pancreatitis: focal pancreatitis or cancer? Is there a role for FNA/biopsy? Autoimmune pancreatitis. Endoscopy. 2006 Jun;38 Suppl 1:S30-5. doi: 10.1055/s-2006-946648. No abstract available. PMID 16802220
- [Result] Levy MJ. Endoscopic ultrasound-guided trucut biopsy of the pancreas: prospects and problems. Pancreatology. 2007;7(2-3):163-6. doi: 10.1159/000104240. Epub 2007 Jun 21. PMID 17592229
- [Result] Suda K, Takase M, Fukumura Y, Ogura K, Ueda A, Matsuda T, Suzuki F. Histopathologic characteristics of autoimmune pancreatitis based on comparison with chronic pancreatitis. Pancreas. 2005 May;30(4):355-8. doi: 10.1097/01.mpa.0000160283.41580.88. PMID 15841047
- [Result] Notohara K, Burgart LJ, Yadav D, Chari S, Smyrk TC. Idiopathic chronic pancreatitis with periductal lymphoplasmacytic infiltration: clinicopathologic features of 35 cases. Am J Surg Pathol. 2003 Aug;27(8):1119-27. doi: 10.1097/00000478-200308000-00009. PMID 12883244
- [Result] Hoshimoto S, Aiura K, Tanaka M, Shito M, Kakefuda T, Sugiura H. Mass-forming type 1 autoimmune pancreatitis mimicking pancreatic cancer. J Dig Dis. 2016 Mar;17(3):202-209. doi: 10.1111/1751-2980.12316. PMID 27121246
- [Result] Weber SM, Cubukcu-Dimopulo O, Palesty JA, Suriawinata A, Klimstra D, Brennan MF, Conlon K. Lymphoplasmacytic sclerosing pancreatitis: inflammatory mimic of pancreatic carcinoma. J Gastrointest Surg. 2003 Jan;7(1):129-37; discussion 137-9. doi: 10.1016/s1091-255x(02)00148-8. PMID 12559194